CLINICAL TRIAL: NCT02793609
Title: Outpatient Versus Inpatient Double Balloon Catheter for Induction of Labor: a Randomised Trial
Brief Title: Outpatient Versus Inpatient Balloon Catheter Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: T169/2016
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Prolonged Pregnancy
Keywords: induction of labor; double balloon catheter; mechanical ripening
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient group (Other): After insertion of double balloon induction catheter of labor, women are discharged overnight to home. Intervention is to let patient to go home.
  Interventions: Other: Intervention is to let patient to go home.
- Inpatient group (Other): After insertion of double balloon induction catheter of labor, women are observed in the prenatal ward. Intervention is to observe women in the ward.
  Interventions: Other: Intervention is to observe women in the ward.

INTERVENTIONS:
Other: Intervention is to let patient to go home. — Intervention is to let patient to go home.
  Arms: Outpatient group
Other: Intervention is to observe women in the ward. — Intervention is to observe women in the ward.
  Arms: Inpatient group

SUMMARY:
Randomized trial comparing double balloon catheter for induction of labor between in- and outpatient groups.Investigators assess feasibility, clinical effectiveness and patient acceptability of outpatient versus inpatient catheter for induction of labor.

DETAILED DESCRIPTION:
The objective of this study is to describe labor outcomes in women with double balloon induction catheter of labor. Participants included are women with uncomplicated singleton pregnancy of ≥37- ≤41+5 weeks of gestation. Patients are randomized to two groups: one hundred are randomized to the inpatient and one hundred to the outpatient group.

The main outcome measure is the pain evaluated by VAS at one, five, nine and 13 hours after the placement of double balloon induction catheter. The total hospital stay and induction to delivery interval time is measured. Also the mode of birth as well as maternal and neonatal morbidity and patient satisfaction are recorded.

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated pregnancy
* singleton pregnancy
* pregnancy weeks between >37 and <41+5
* the patient is living in 1/2 hour away from hospital

Exclusion Criteria:

* patient has any disease or medication
* multiple pregnancy
* pregnancy week > 41+5
* preterm rupture of membranes
* patient living more than 1/2 hour away from hospital

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The pain measured by visual analogy scale(VAS) after double balloon catheter | During the induction of the labor and postpartum period in the hospital.
  Visual analogy score assessed by patient. Minimum 1mm to maximum 100 mm.

SECONDARY OUTCOMES:
The maternal morbidity | during the induction of the labor and postpartum period in the hospital
  number of mothers having any kind of infection
The total hospital stay in both groups | maximum 14 days
  length in days
neonatal morbidity | during the induction of the labor and postpartum period in the hospital
  number of babies having any kind of infection

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi M Rinne, PhD, Principal Investigator — Turku University Hospital; Päivi ML Polo, PhD, Study Director — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided
Letter to patients.

REFERENCES:
- [Background] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Background] Prager M, Eneroth-Grimfors E, Edlund M, Marions L. A randomised controlled trial of intravaginal dinoprostone, intravaginal misoprostol and transcervical balloon catheter for labour induction. BJOG. 2008 Oct;115(11):1443-50. doi: 10.1111/j.1471-0528.2008.01843.x. Epub 2008 Aug 19. PMID 18715244
- [Result] Henry A, Madan A, Reid R, Tracy SK, Austin K, Welsh A, Challis D. Outpatient Foley catheter versus inpatient prostaglandin E2 gel for induction of labour: a randomised trial. BMC Pregnancy Childbirth. 2013 Jan 29;13:25. doi: 10.1186/1471-2393-13-25. PMID 23356673
- [Derived] Alfirevic Z, Gyte GM, Nogueira Pileggi V, Plachcinski R, Osoti AO, Finucane EM. Home versus inpatient induction of labour for improving birth outcomes. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007372. doi: 10.1002/14651858.CD007372.pub4. PMID 32852803